CLINICAL TRIAL: NCT02650427
Title: A Pilot Study to Evaluate the Safety of a 3 Weeks Sitagliptin Treatment in HCC Patients Undergoing Liver Resection
Acronym: HCC-DPPIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C15-41; 2015-002968-17 (EudraCT Number)
Record Dates: First submitted 2015-12-22; First posted 2016-01-08 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2018-10

CONDITIONS: Hepato Carcinoma
MeSH Terms: interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DPPIV Inhibition (Experimental): The study will include 3 weeks administration (± 7 days) of sitagliptin as monotherapy (taken orally). The study will use 3 doses: the first five patients will receive 100 mg/day, the next five 200 mg/day and the last five patients 600 mg/day. During this time, arrangements will be made for surgical resection, as per the standard of care treatment of patients. Blood samples will be obtained for immunology studies. The study will end one week after surgery. Patients will continue their treatment for HCC as prescribed by the clinician.
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — 100mg or 200mg or 600mg, daily for 3 weeks ± 7 days
  Other Names: Januvia

SUMMARY:
Boosting of tumor cell killing by cytotoxic lymphocytes may be a promising means to enhance anti-tumor immunity. Prior studies demonstrated that tumor infiltration by cytotoxic lymphocytes correlates with control of tumor growth and is associated with an improved prognosis in cancer patients. Trafficking of activated lymphocytes is a tightly regulated mechanism and the specific nature of the chemokine milieu is a crucial determinant for permitting T cell entry into the tumor microenvironment. CXCL10 is an interferon-inducible chemokine particularly important for the recruitment of activated T, and it has been shown to enhance anti-tumor responses through its action on cytotoxic T cells (e.g., glioblastoma, colorectal adenocarcinoma and lung carcinoma). Additionally, roles for CXCL10 as an anti-tumor effector include its ability to chemo-attract NK cells into sites of inflammation, and its ability to inhibit development of new vasculature and induce the regression of newly formed vessels. Adding a layer of complexity, the function of CXCL10 can be regulated by dipeptidylpeptidase IV (DPPIV), leading to the formation of a dominant negative, antagonist form of the chemokine. This was initially demonstrated in vitro, and recent work has provided convincing in vivo evidence that antagonist forms of CXCL10 regulate lymphocyte trafficking. The main goal of this protocol is to evaluate the tolerance of sitagliptin treatment in HCC patients, and secondary DPPIV inhibitors as a strategy for protecting CXCL10 chemokine agonist activity as a means to enhance tumor regression.

DETAILED DESCRIPTION:
The study will be conducted in 15 patients. Patient selection will be made based on medical records during a weekly staff meeting. After collection of informed consent, the patients will undergo a biopsy of the tumor and of the not-tumoral liver and 2-4 weeks later HCC resection.

The study will include a phase of 3 weeks [± 7 days] administration of sitagliptin as monotherapy (taken orally) after liver biopsy and before HCC resection. The window of ± 7 days is deliberately wide to take in account the variable arrangements made for surgical resection. Nevertheless we will make our efforts to focus on a three weeks regimen. Three doses of sitagliptin will be used: 1) 100mg/day (dose recommended in the SmCP), 2) 200mg/day and 3) 600mg/day; with 5 patients in each group. Arrangements will be made for surgical resection upon standard care. Blood samples will be obtained for immunology studies at each visit. The study will end one week after surgery (or less if the state of health of the patient does not require to stay longer in the hospital). Patients will continue their treatment for HCC as prescribed by the clinician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years old the day of inclusion.
* For women, a negative blood pregnancy test before inclusion is necessary. Note: this test will be done only to women of childbearing age and non menopausal.
* HCC based on medical imaging with indication of liver resection and without contra-indication of preoperative liver biopsy.
* Minor resection not exceeding 2 liver segments
* No cirrhosis or cirrhosis with a Child-Pugh Score Class A. Note: this score is used worldwide to assess liver function in cirrhosis.
* Informed consent must be obtained for all subjects prior to study entry.
* Patients affiliated to health policy insurance.

Exclusion Criteria:

* Presence of HIV Infection.
* Presence of renal impairment (CrCl <60 ml / min).
* Liver function compromised (Child Pugh B, MELD score > 9)
* Indirect sign of portal hypertension (Oesophagal Varices, splenomegaly, platelet count less than 100.000)
* A need for major hepatic resection (more than 2 segments)
* Taking digoxin (digitalis) within 6 months of starting treatment.
* History of severe hypersensitivity reaction (such as anaphylactic shock or angioedema) to sitagliptin.
* Patients with diabetes.
* Pregnant or absence of an effective contraception for women.
* A person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure.
* Living conditions suggesting an inability to track all scheduled visits by the protocol.
* Life expectancy less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Safety (Number of adverse events. Toxicity grade > 3) | After Day 0 until the end of the trial, i.e. a duration of 3 weeks +/- 7 days for each patient

SECONDARY OUTCOMES:
DPPIV Activity | Baseline; week 1, 3 of sitagliptin therapy , 3 days after end of sitagliptin therapy
  Plasma concentration and activity of DPPIV (measured using an ELISA and a luciferase bioassay, respectively).
CXCL10 truncation | Baseline; week 1, 3 of sitgaliptin therapy, 3 days after end of sitagliptin therapy
  Monitoring the short and the long form of IP-10 as compared to the total plasma concentration (three distinct ELISA assays).
Immune cells trafficking | Baseline; week 1, 3 of sitagliptin therapy, 3 days after end of sitagliptin therapy
  Frequency of CXCR3+ cells in circulation (monitored by FACS).
Infiltration of leucocytes in tumor tissue | Baseline, week 3 of sitagliptin therapy
  Histochemical method with a panel of Ab.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier SCATTON, Principal Investigator — Pitié-Salpêtrière Hospital, Paris, France
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This paper reports results of this study — https://pasteur.hal.science/pasteur-03384283v1/file/Safety_of_sitagliptin_in_treatment_of_hepatocellul.pdf